CLINICAL TRIAL: NCT03754101
Title: Exome Sequencing Study in Cardiomyopathy to Identify New Risk Variants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Dao Wen Wang, Professor, Tongji Hospital
Other Study IDs: TJ-DM-GENE
Record Dates: First submitted 2018-11-01; First posted 2018-11-27 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Genetic mutations has been proved to be associated wth the onset of cardiomyopathy. In the present study, we intend to identify new related variants or genes. From March, 2003 to November, 2017, patients diagnosed as cardiomyopathy were consecutively recruited, and their sampled were drawn from peripheral blood. Paired control group were also enrolled. The whole exome sequencing was used to find out the variants associated with the onset of cardiomyopathy and its prognosis.

ELIGIBILITY:
Inclusion Criteria:

· Patients diagnosed as cardiomyopathy according to the definition of American Heart Association

Exclusion Criteria:

* Uncontrolled hypertension significant valvular disease
* Mild ischemic heart disease
* Significant systemic infection
* Thyroid-induced cardiomyopathy
* Excessive alcohol consumption
* Precious cancer treatment including irradiation
* Refusal to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: hospitalized patients with cardiomyopathy will be enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2003-03-03 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular death confirmed by death comfirmation or interview with the relatives | up to 24 months
  Death from cardiovascular causes and any unknown death unless there was another certain cause
Heart transplantation confirmed by medical record | up to 24 months
  Heart transplantation within 24 months

SECONDARY OUTCOMES:
All cause death confirmed by death comfirmation or interview with the relatives | up to 24 months
  Any death at hospital or after discharge
Heart failure recurring confirmed by medical record | up to 24 months
  Recurrence of heart failure at hospital or after discharge

OTHER OUTCOMES:
Readmission because of cardiovascular diseases confirmed by medical record | up to 24 months
  Readmission because of cardiovascular diseases within 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Dao Wen Wang, Doctor, Study Chair — Tongji Hospital,Wuhan, Hubei, China, 430030
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li S, Sun Y, Hu S, Hu D, Li C, Xiao L, Chen Y, Li H, Cui G, Wang DW. Genetic risk scores to predict the prognosis of chronic heart failure patients in Chinese Han. J Cell Mol Med. 2020 Jan;24(1):285-293. doi: 10.1111/jcmm.14722. Epub 2019 Oct 31. PMID 31670483